CLINICAL TRIAL: NCT06494462
Title: Effect of Gamification-Based Virtual Reality Application and Video-Assisted Teaching Methods on Nursing Students' Skill Learning and Confidence Levels in Subcutaneous Injection Training
Brief Title: Gamification-Based Virtual Reality in Subcutaneous Injection Skill Teaching
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Nihal Taskiran, Principal Investigator, Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Adnan Menderes Univ-Nursing
Record Dates: First submitted 2024-06-20; First posted 2024-07-10 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2024-10

CONDITIONS: Training Group
Keywords: virtual reality; game; subcutaneous injection; skill; nursing students; confidence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- game based virtual reality (Experimental): 24 hours after the theoretical lecture, students will be given a demonstrative presentation of the application in the laboratory environment by the instructor (researcher).
  All students will perform the application on low-fidelity models (task trainers) under the supervision of the instructor.
  After the laboratory application, students will be required to play a gamified virtual reality experience using Oculus 2 Interactive Virtual Reality Headsets within 7 days before the clinical application.
  Interventions: Other: virtual reality training
- Video (Experimental): 24 hours after the theoretical lecture, students will be given a demonstrative presentation of the application in the laboratory environment by the instructor (researcher).
  All students will perform the application on low-fidelity models (task trainers) under the supervision of the instructor.
  After the laboratory application, students will be shown a video recording prepared by the researchers via VR Box non-interactive virtual reality headsets within 7 days before the clinical application.
  Interventions: Other: virtual reality training
- Control (No Intervention): 24 hours after the theoretical lecture, students will be given a demonstrative presentation of the application in the laboratory environment by the instructor (researcher).
  All students will perform the application on low-fidelity models (task trainers) under the supervision of the instructor.

INTERVENTIONS:
Other: virtual reality training — students will watch a video about subcutaneous injection or students will play a about subcutaneous injection by virtual reality glasses
  Arms: Video; game based virtual reality

SUMMARY:
This randomized controlled experimental study aimed to determine the effect of gamification-based virtual reality applications and video demonstration methods on nursing students' skill learning and confidence levels in subcutaneous injection skill training.

The population of the study consisted of 96 first-year nursing students enrolled in the Fundamentals of Nursing course at a university's Faculty of Nursing during the spring semester of the 2024-2025 academic year. The students will be randomized into three groups, each containing 32 students: two experimental groups and one control group. First, the topic of subcutaneous injection application will be theoretically explained to all students for 90 minutes. After completing the theoretical explanation, the skill of subcutaneous injection application will be taught in a laboratory setting using the Gamification-Based Virtual Reality Application + Demonstration method for students in Experimental Group 1, the Video Demonstration + Demonstration method for students in Experimental Group 2, and only the Demonstration method for students in the Control Group. After the theoretical explanation and laboratory practices according to their groups, the subcutaneous injection skill levels of the students in all three groups will first be assessed in the laboratory setting using the Objective Structured Clinical Examination (OSCE) and later evaluated in the clinical setting using the Subcutaneous Injection Skill Checklist. The confidence levels of the students will be determined through self-reporting using the "Confidence Scale" after all clinical practices are completed.

The research data will be collected between April and June 2025. Descriptive (number, percentage, mean, standard deviation, minimum-maximum) and comparative statistics (Chi-Square Test, Mann Whitney U Test, Wilcoxon Test) will be used in the analysis of the data. The level of statistically significance will be considered at p<0.05.

DETAILED DESCRIPTION:
Nursing education is a structured educational system designed to impart a professional nursing identity to students and prepare them for professional life. This system integrates theoretical and practical education as a whole. It aims to develop cognitive, affective, and psychomotor skills, as well as critical thinking, decision-making, and problem-solving abilities.

The primary objective is to determine the most effective learning method by comparing two different methods in teaching the subcutaneous injection skill, one of the most frequently encountered invasive procedures in clinical practice. The secondary objective is to assess the impact of the applied learning methods on students' confidence levels. Additionally, it aims to demonstrate the usability and effectiveness of these methods in nursing skill education.

The population of the research will consist of first-year nursing students (N=280) enrolled in the Fundamentals of Nursing course at the Faculty of Nursing of a university in the spring semester of the 2024-2025 academic year.The "G. Power-3.1.9.2" program was used to estimate the appropriate number of students needed for a study sample. It was found through power analysis that a sample size of 96 students (p<0.05 significance) provided an 88% theoretical power with 95% confidence and 0.30 effect size. The students to be sampled will be randomly selected from the population using the simple random sampling method, considering a random number table, and will be equally divided into Experiment-1 (n=32), Experiment-2 (n=32), and Control (n=32) groups.

The subject of subcutaneous injection, which is planned to be taught within the scope of the research, will be explained theoretically to all students face-to-face in the classroom environment for 2 class hours (90 min), and then the students will be made to practice the skill on low-reality models in the laboratory for 4 class hours (180 min). In the laboratory, subcutaneous injection skill will be shown to all students by the researchers by demonstration method and students will be ensured to repeat the application until they learn the skill.

"Student Information Form", "SC Injection Skill Checklist", "Self-Confidence Scale" will be used in collecting research data.

Student Information Form: It consists of 8 questions characteristics of the students such as age, gender, graduated high school, city of residence for the longest time, desire for nursing profession and reason for choosing the profession, technology usage status.

SC Injection Skill Checklist: The form prepared by the researchers in line with the literature information was prepared to measure the skill levels of the students regarding SC injection. The prepared form will be sent to 3 faculty members who are experts in the field of Fundamentals of Nursing and who have studies on SC injection and expert opinion will be obtained before the start of the study to be evaluated for suitability. The form consisting of 27 items in which each application step is scored shows the skill level as a score.

Self-confidence Scale (SCS): Self-confidence scale developed by Akın (2007) by adopting self-efficacy theory within the scope of Bandura's social-cognitive theory consists of 33 items collected under two factors as internal self-confidence and external self-confidence. In the self-report and 5-point Likert-type scale, 17 items collected under the internal self-confidence factor are mostly related to individuals' self-confidence towards themselves, while the external self-confidence dimension consisting of 16 items is related to individuals' self-confidence towards their external environment and social life. The internal consistency reliability coefficients of the scale are 0.91 for the whole scale, 0.83 for the internal self-confidence dimension and 0.85 for the external self-confidence dimension.

After the theoretical and laboratory applications are completed according to their respective groups, the skill learning levels of students in all three groups will be evaluated by Objective Structured Clinical Examination (OSCE) in laboratory and Subcutaneous Injection Skill Checklist in clinics of the University Hospital.

Finally, in the last week of the clinical application, the confidence levels of students in all three groups will be evaluated using the "Confidence Scale".

Statistical Analysis of Data The data obtained from the research will be analyzed using the IBM SPSS (Statistical Package for Social Science) 25.0 software. Descriptive statistics (number, percentage, mean, standard deviation, minimum-maximum) and comparative statistics (Chi-Square Test, Mann Whitney U Test, Wilcoxon Test) will be used in the analysis of the data. A p-value of less than 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* To be between 18-50 years old
* To be a student of nursing department
* Being a 1st year nursing student
* To volunteer to participate in the research
* Having internet access

Exclusion Criteria:

* Being a graduate of a of health vocational high school
* Having received training on SC injection,
* Have a clinical experience,
* To be absent from the theoretical and laboratory courses on the dates of SC injection subject

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2024-01-07 (Actual); Primary Completion 2025-06-02 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
Skill Evaluation | twice, first evaluation will take place up to 10 weeks after the begining of the study (end of laboratory training) and second evaluation will take place up to 12 weeks the begining of the study (after 7 or 15 days the laboratory training) in hospital
  First, the evaluation will be conducted using the Objective Structured Clinical Examination (OSCE).The OSCE score will be determined according to the procedure steps specified in the SC Injection Skill Checklist. The form consisting of 27 items in which each application step is scored shows the skill level as points. In the evaluation, each step that the student performs correctly will be calculated as 2 points, each incomplete step will be calculated as 1 point, and each step that the student does not perform or performs incorrectly will be calculated as 0 points. The lowest score that can be obtained from the form is 0 and the highest score is 54.
  In the second stage, all students will be evaluated in Clinics of the University Hospital. Skill assessments will be performed using the Subcutaneous Injection Skill Checklist.The average score obtained as a result of the two assessments will determine the student's skill level.

SECONDARY OUTCOMES:
Confidence | once, up to 20 weeks (when the research is finished)
  The confidence levels of students in all three groups will be evaluated using the " Self Confidence Scale". The scale consists of 33 items collected under two factors as internal self-confidence and external self-confidence. In the self-report and 5-point Likert-type scale, 17 items collected under the internal self-confidence factor are mostly related to individuals' self-confidence towards themselves, while the external self-confidence dimension consisting of 16 items is related to individuals' self-confidence towards their external environment and social life. The highest score that can be obtained from the scale is 165 and the lowest score is 33. A high score obtained from the scale indicates a high level of self-confidence. The total score obtained from the scale divided by the number of items determines the level of self-confidence. Accordingly, <2.5 indicates low self-confidence, 2.5-3.5 indicates medium self-confidence, and 3.5 and above indicates high self-confidence.

CONTACTS AND LOCATIONS:
Overall Officials: Barış Atiker, Principal Investigator — Aydin Adnan Menderes University
Locations (1):
- Adnan Menderes University Nursing Faculty, Aydin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The data that support the findings of this study are available onrequest from the corresponding author.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: end of the study
Access Criteria: The data that support the findings of this study are available onrequest from the corresponding author.